CLINICAL TRIAL: NCT01474239
Title: Randomized Non Comparative Phase II Trial With Bevacizumab and Fotemustine in the Treatment of Recurrent Glioblastoma
Brief Title: A Study of Avastin (Bevacizumab) And Fotemustine in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML25739
Record Dates: First submitted 2011-11-08; First posted 2011-11-18 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2015-09

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; fotemustine

ARMS (2):
- Calibration Arm (Experimental)
  Interventions: Drug: fotemustine
- Investigational Arm (Experimental)
  Interventions: Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 10 mg/kg every 2 weeks intravenously until disease progression or unacceptable toxicity
  Arms: Investigational Arm
Drug: fotemustine — 75 mg/m2 intravenously on days 1, 8 and 15 followed by, after a 5 weeks interval, 100 mg/m2 on day 1 of a 3-weeks cycle. Until disease progression or unacceptable toxicity
  Arms: Calibration Arm

SUMMARY:
This randomized, non-comparative study will evaluate the efficacy and safety of Avastin (bevacizumab) in patients with recurrent glioblastoma. Patients will be randomized to receive Avastin 10 mg/kg intravenously every 2 weeks or fotemustine 75 mg/m2 on days 1, 8 and 15, followed by, after a 5 weeks interval, 100 mg/m2 intravenously every 3 weeks. Treatment with fotemustine serves as a calibration arm and no formal efficacy comparison will be made between the two treatment arms. The anticipated time of study treatment is until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/=18 years of age
* Diagnosis of recurrent glioblastoma multiforme (Grade IV)
* Previous treatment with temozolomide and radiotherapy
* First recurrence after standard adjuvant treatment (surgery, followed by radiotherapy and chemotherapy)
* Adequate hematological, biochemical and organ functions

Exclusion Criteria:

* Previous treatment with Avastin or other anti-angiogenic drugs
* Residual relevant toxicity resulting from previous therapy
* Radiotherapy within the 3 months prior to the diagnosis of disease progression
* Chemotherapy in the previous 4 weeks
* Other active or inactive malignancies (except for carcinoma in situ of the cervix, of the prostate or basal cell carcinoma)
* Clinically significant cardiovascular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2011-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Italy (9):
  - San Giovanni Rotondo, Apulia
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Terni, Umbria
  - Padua, Veneto
  - Treviso, Veneto

REFERENCES:
- [Derived] Brandes AA, Finocchiaro G, Zagonel V, Reni M, Caserta C, Fabi A, Clavarezza M, Maiello E, Eoli M, Lombardi G, Monteforte M, Proietti E, Agati R, Eusebi V, Franceschi E. AVAREG: a phase II, randomized, noncomparative study of fotemustine or bevacizumab for patients with recurrent glioblastoma. Neuro Oncol. 2016 Sep;18(9):1304-12. doi: 10.1093/neuonc/now035. Epub 2016 Mar 6. PMID 26951379

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study included 28-day screening period. Participants were randomized according to a 2:1 ratio to one of the 2 treatment groups. A total of 99 participants were screened, of which 91 were randomized.
Groups:
- Bevacizumab: Participants received bevacizumab 10 milligrams per kilogram (mg/kg) via intravenous (IV) infusion every 14 days until disease progression was radiographically documented or the onset of toxicity prevented treatment continuation.
- Fotemustine: Participants received fotemustine 75 milligrams per square meter (mg/m^2) via IV infusion on Days 1, 8, and 15 (induction phase), followed by a 35-day drug-free interval, and then fotemustine 100 mg/m^2 every 21 days (maintenance phase) until disease progression was radiographically documented or the onset of toxicity prevented treatment continuation.
Period: Overall Study
Arm/Group | Bevacizumab | Fotemustine
Started | 59 | 32
Completed | 0 | 0
Not Completed | 59 | 32
Not completed — Disease Progression | 37 | 25
Not completed — Adverse Event | 12 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 1 | 1
Not completed — Clinical Disease Progression | 7 | 1
Not completed — Withdrawal for Economic Reason | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants with at least one administration of the study drug and at least one safety assessment.
Groups:
- Bevacizumab: Participants received bevacizumab 10 mg/kg via IV infusion every 14 days until disease progression was radiographically documented or the onset of toxicity prevented treatment continuation.
- Fotemustine: Participants received fotemustine 75 mg/m^2 via IV infusion on Days 1, 8, and 15 (induction phase), followed by a 35-day drug-free interval, and then fotemustine 100 mg/m^2 every 21 days (maintenance phase) until disease progression was radiographically documented or the onset of toxicity prevented treatment continuation.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Fotemustine | Total
Number analyzed (Participants) | 59 | 32 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.86 (9.40) | 55.63 (10.64) | 56.43 (9.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 9 | 29
  Male | 39 | 23 | 62

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Alive 6 Months After Start of Treatment
Description: Overall survival (OS) was defined as the time in months from the start of treatment to death due to any cause. If a participant was not known to have died, time was censored at the last date the participant was known to be alive, which was defined as the latest among date of last visit, date of last sample collected for laboratory exam, date of magnetic resonance imaging (MRI) assessment, date of last treatment, date of discontinuation and date of last available follow-up visit. Participants with no information after baseline were censored at Day 1. OS was estimated by the Kaplan-Meier method.
Time Frame: 6 months
Population: Intent-to-Treat (ITT) population included all randomized participants with at least one administration of the study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
percentage of participants | 62.07 [48.37 to 74.49] | 73.33 [54.11 to 87.72]
Statistical Analysis 1: Comparison: Bevacizumab; The 6-month OS rate (OS-6) for bevacizumab was compared to the expected proportion of 0.60 under null hypothesis (ineffective treatment) with the application of the exact binomial test. The one-tailed statistical hypotheses was p0 less than or equal to (≤) 0.60 (null hypothesis) versus pA greater than or equal to (≥) 0.77 (alternative hypothesis), where p is the estimated probability of survival at 6 months; Test type: Superiority or Other; p = 0.4291, Exact Binomial Test — Statistical significance was assessed with a one-sided alpha error of 10 percent (%)

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time in months from the start of treatment to death due to any cause. If a participant was not known to have died, time was censored at the last date the participant was known to be alive, which was defined as the latest among date of last visit, date of last sample collected for laboratory exam, date of MRI assessment, date of last treatment, date of discontinuation and date of last available follow-up visit. Participants with no information after baseline were censored at Day 1. OS was estimated by the Kaplan-Meier method.
Time Frame: Baseline until death (up to 691 days)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
months | 7.26 [5.82 to 9.20] | 8.66 [6.34 to 15.38]

3. Secondary Outcome: Percentage of Participants Who Were Alive and Progression Free 6 Months After Start of Treatment
Description: Progression-free survival (PFS) was defined as the time in months from the start of treatment to the date of the first occurrence of disease progression or death from any cause, whichever occurred first. PFS was estimated by the Kaplan-Meier method. Progression was assessed using Response Assessment in Neuro-Oncology (RANO) or Macdonald Response Criteria, whichever occurred first. As per the RANO criteria, progression was defined as 25% or more increase in enhancing lesions despite stable or increasing steroid dose; increase (significant) in non-enhancing T2/FLAIR lesions, not attributable to other non-tumor causes; any new lesions; and clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease). As per the Macdonald criteria, progression was defined as 25% or more increase in enhancing lesions; any new lesions; and clinical deterioration.
Time Frame: 6 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
percentage of participants | 26.32 [15.54 to 39.66] | 10.71 [2.27 to 28.23]

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time in months from the start of treatment to the date of the first occurrence of disease progression or death from any cause, whichever occurred first. PFS was estimated by the Kaplan-Meier method. Progression was assessed using the RANO or the Macdonald Response Criteria, whichever occurred first. As per RANO criteria, progression was defined as 25% or more increase in enhancing lesions despite stable or increasing steroid dose; increase (significant) in non-enhancing T2/FLAIR lesions, not attributable to other non-tumor causes; any new lesions; and clinical deterioration (not attributable to other non-tumor causes and not due to steroid decrease). As per Macdonald criteria, progression was defined as 25% or more increase in enhancing lesions; any new lesions; and clinical deterioration.
Time Frame: Baseline until disease progression or death (baseline, 46 days after first administration of study drug, and thereafter every 56 days up to 691 days)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
months | 3.38 [3.15 to 4.37] | 3.45 [1.87 to 3.84]

5. Secondary Outcome: Percentage of Participants Alive 9 Months After Start of Treatment
Description: as for outcome 2
Time Frame: 9 months
Population: ITT population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
percentage of participants | 37.93 [25.51 to 51.63] | 46.67 [28.34 to 65.67]

6. Secondary Outcome: Percentage of Participants Alive 12 Months After Start of Treatment
Description: as for outcome 2
Time Frame: 12 months
Population: ITT population. Here, the number of participants analyzed signified participants with evaluable data for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 58 | 30
percentage of participants | 25.86 [15.26 to 39.04] | 40.00 [22.66 to 59.40]

7. Secondary Outcome: Percentage of Participants Alive 30 Days After Last Dose of Study Drug
Description: as for outcome 2
Time Frame: 30 days after last dose of study drug (up to Day 600)
Population: ITT population. Here, the number of participants analyzed signified participants with evaluable data for this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 58 | 30
percentage of participants | 93.10 [83.27 to 98.09] | 90.00 [73.47 to 97.89]

8. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR)
Description: Percentage of participants achieving CR or PR as overall response between first drug administration and documented disease progression were calculated. Tumor response was evaluated according to both the RANO and the Macdonald response criteria. As per Macdonald criteria, CR was defined as the disappearance of all enhancing disease, sustained for at least 4 weeks, and no new lesions along with clinical features of clinically stable or improved, with no corticosteroid; PR was defined as a 50% or more decrease of all measurable enhancing lesions, sustained for at least 4 weeks, and no new lesion along with clinical features of clinically stable or improved, with stable or reduced corticosteroids. RANO criteria defined CR and PR the same as Macdonald criteria with the following additions: CR - improved non enhancing T2/FLAIR lesions; PR - no progression of non-measurable disease, stable or improved non enhancing FLAIR/T2 lesions.
Time Frame: as for outcome 4
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
percentage of participants
  RANO Evaluation | 28.81 | 9.38
  MacDonald Evaluation | 28.81 | 6.25

9. Secondary Outcome: Change From Screening in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) Scores at Weeks 8, 16, 24, 32, 40, 48, 56, 64, and 72
Description: EORTC QLQ-C30: included global health status/quality of life (QOL), functional scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Most questions used a 4-point scale (1 'Not at All' to 4 'Very Much'); 2 questions used a 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores were averaged and transformed to 0-100 scale; a higher score for Global QOL/functional scales indicates better level of QOL/functioning, or a higher score for symptom scale indicates greater degree of symptoms.
Time Frame: Screening, Weeks 8, 16, 24, 32, 40, 48, 56, 64, and 72
Population: ITT population. Here, the number of participants analyzed signified participants with evaluable data for this outcome, and "n" signified participants with evaluable data for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 58 | 31
units on a scale
  Physical Functioning (Fn): Screening (n=58,31) | 71.95 (25.65) | 78.92 (25.07)
  Physical Fn: Change at Week 8 (n=27,16) | 10.37 (19.07) | 7.08 (12.76)
  Physical Fn: Change at Week 16 (n=15,7) | 7.56 (19.17) | 8.57 (13.72)
  Physical Fn: Change at Week 24 (n=14,1) | 13.81 (24.17) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Physical Fn: Change at Week 32 (n=7,2) | 18.10 (28.21) | 13.33 (9.43)
  Physical Fn: Change at Week 40 (n=9,1) | 4.44 (19.72) | 6.67 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Physical Fn: Change at Week 48 (n=4,1) | 3.33 (16.78) | 6.67 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Physical Fn: Change at Week 56 (n=4,0) | 6.67 (9.43) | NA (NA) — Data not available as no participant was evaluable.
  Physical Fn: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Physical Fn: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Role Fn: Screening (n=58,31) | 67.82 (31.04) | 73.66 (32.14)
  Role Fn: Change at Week 8 (n=27,16) | 6.17 (34.01) | 4.17 (21.52)
  Role Fn: Change at Week 16 (n=15,7) | 2.22 (25.87) | 2.38 (26.23)
  Role Fn: Change at Week 24 (n=14,1) | 14.29 (33.88) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Role Fn: Change at Week 32 (n=7,2) | 16.67 (28.87) | 0.00 (0.00)
  Role Fn: Change at Week 40 (n=9,1) | 0.00 (22.05) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Role Fn: Change at Week 48 (n=4,1) | 0.00 (36.00) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Role Fn: Change at Week 56 (n=4,0) | -12.50 (36.96) | NA (NA) — Data not available as no participant was evaluable.
  Role Fn: Change at Week 64 (n=1,0) | -50.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Role Fn: Change at Week 72 (n=1,0) | -50.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Emotional Fn: Screening (n=58,31) | 73.56 (23.47) | 74.19 (23.41)
  Emotional Fn: Change at Week 8 (n=27,16) | -8.02 (23.62) | 8.33 (24.91)
  Emotional Fn: Change at Week 16 (n=15,7) | -0.56 (14.25) | -2.38 (27.52)
  Emotional Fn: Change at Week 24 (n=14,1) | 10.12 (29.63) | -33.33 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Emotional Fn: Change at Week 32 (n=7,2) | -2.38 (15.00) | 16.67 (0.00)
  Emotional Fn: Change at Week 40 (n=9,1) | -5.56 (24.65) | 8.33 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Emotional Fn: Change at Week 48 (n=4,1) | 14.58 (27.53) | 8.33 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Emotional Fn: Change at Week 56 (n=4,0) | -4.17 (27.64) | NA (NA) — Data not available as no participant was evaluable.
  Emotional Fn: Change at Week 64 (n=1,0) | 8.33 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Emotional Fn: Change at Week 72 (n=1,0) | 8.33 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Cognitive Fn: Screening (n=58,31) | 70.40 (25.18) | 79.03 (24.33)
  Cognitive Fn: Change at Week 8 (n=27,16) | 4.94 (23.49) | 7.29 (23.55)
  Cognitive Fn: Change at Week 16 (n=15,7) | 2.22 (17.67) | -4.76 (34.31)
  Cognitive Fn: Change at Week 24 (n=14,1) | 10.71 (24.11) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Cognitive Fn: Change at Week 32 (n=7,2) | 0.00 (16.67) | 8.33 (11.79)
  Cognitive Fn: Change at Week 40 (n=9,1) | -1.85 (19.44) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Cognitive Fn: Change at Week 48 (n=4,1) | 0.00 (0.00) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Cognitive Fn: Change at Week 56 (n=4,0) | -4.17 (20.97) | NA (NA) — Data not available as no participant was evaluable.
  Cognitive Fn: Change at Week 64 (n=1,0) | 16.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Cognitive Fn: Change at Week 72 (n=1,0) | 16.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Social Fn: Screening (n=58,31) | 72.99 (28.07) | 81.18 (24.24)
  Social Fn: Change at Week 8 (n=27,16) | 1.85 (31.12) | 4.17 (23.96)
  Social Fn: Change at Week 16 (n=15,7) | 1.11 (27.07) | -2.38 (26.23)
  Social Fn: Change at Week 24 (n=14,1) | 13.10 (39.32) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Social Fn: Change at Week 32 (n=7,2) | -7.14 (38.32) | 8.33 (11.79)
  Social Fn: Change at Week 40 (n=9,1) | -5.56 (22.05) | 16.67 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Social Fn: Change at Week 48 (n=4,1) | -4.17 (36.96) | 16.67 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Social Fn: Change at Week 56 (n=4,0) | -12.50 (28.46) | NA (NA) — Data not available as no participant was evaluable.
  Social Fn: Change at Week 64 (n=1,0) | -66.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Social Fn: Change at Week 72 (n=1,0) | -66.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  QOL: Screening (n=58,31) | 58.05 (26.40) | 66.13 (24.90)
  QOL: Change at Week 8 (n=27,16) | -3.09 (20.17) | 6.25 (22.87)
  QOL: Change at Week 16 (n=15,7) | -4.44 (14.39) | 7.14 (23.78)
  QOL: Change at Week 24 (n=14,1) | 4.76 (21.11) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  QOL: Change at Week 32 (n=7,2) | 3.57 (17.91) | -12.50 (17.68)
  QOL: Change at Week 40 (n=9,1) | -2.78 (25.34) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  QOL: Change at Week 48 (n=4,1) | 10.42 (14.23) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  QOL: Change at Week 56 (n=4,0) | 2.08 (34.94) | NA (NA) — Data not available as no participant was evaluable.
  QOL: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  QOL: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Fatigue: Screening (n=58,31) | 31.99 (25.50) | 24.01 (22.05)
  Fatigue: Change at Week 8 (n=27,16) | -3.29 (32.59) | -13.19 (25.73)
  Fatigue: Change at Week 16 (n=15,7) | 2.22 (21.50) | -9.52 (17.48)
  Fatigue: Change at Week 24 (n=14,1) | -6.35 (29.79) | -11.11 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Fatigue: Change at Week 32 (n=7,2) | 3.17 (17.82) | -5.56 (7.86)
  Fatigue: Change at Week 40 (n=9,1) | 9.88 (23.20) | -11.11 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Fatigue: Change at Week 48 (n=4,1) | -8.33 (18.98) | -11.11 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Fatigue: Change at Week 56 (n=4,0) | 2.78 (30.60) | NA (NA) — Data not available as no participant was evaluable.
  Fatigue: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Fatigue: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Nausea: Screening (n=58,31) | 2.01 (7.70) | 1.08 (4.16)
  Nausea: Change at Week 8 (n=27,16) | 1.85 (10.68) | -8.33 (14.91)
  Nausea: Change at Week 16 (n=15,7) | 0.00 (6.30) | -14.29 (20.25)
  Nausea: Change at Week 24 (n=14,1) | -5.95 (10.56) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Nausea: Change at Week 32 (n=7,2) | -2.38 (6.30) | 0.00 (0.00)
  Nausea: Change at Week 40 (n=9,1) | -9.26 (8.78) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Nausea: Change at Week 48 (n=4,1) | 0.00 (0.00) | -16.67 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Nausea: Change at Week 56 (n=4,0) | -4.17 (8.33) | NA (NA) — Data not available as no participant was evaluable.
  Nausea: Change at Week 64 (n=1,0) | -16.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Nausea: Change at Week 72 (n=1,0) | -16.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Pain: Screening (n=58,31) | 6.90 (16.82) | 14.52 (23.47)
  Pain: Change at Week 8 (n=27,16) | -1.85 (24.61) | -6.25 (26.44)
  Pain: Change at Week 16 (n=15,7) | -10.00 (19.72) | -2.38 (20.25)
  Pain: Change at Week 24 (n=14,1) | -8.33 (28.31) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Pain: Change at Week 32 (n=7,2) | 0.00 (16.67) | -8.33 (11.79)
  Pain: Change at Week 40 (n=9,1) | -7.41 (18.84) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Pain: Change at Week 48 (n=4,1) | -29.17 (28.46) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Pain: Change at Week 56 (n=4,0) | 0.00 (19.25) | NA (NA) — Data not available as no participant was evaluable.
  Pain: Change at Week 64 (n=1,0) | -16.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Pain: Change at Week 72 (n=1,0) | -16.67 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Dyspnea: Screening (n=58,31) | 11.49 (22.12) | 3.23 (10.02)
  Dyspnea: Change at Week 8 (n=27,16) | 4.94 (28.80) | -6.25 (21.84)
  Dyspnea: Change at Week 16 (n=15,7) | 0.00 (25.20) | 4.76 (12.60)
  Dyspnea: Change at Week 24 (n=14,1) | -9.52 (27.51) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Dyspnea: Change at Week 32 (n=7,2) | 0.00 (27.22) | 0.00 (0.00)
  Dyspnea: Change at Week 40 (n=9,1) | 3.70 (20.03) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Dyspnea: Change at Week 48 (n=4,1) | -8.33 (16.67) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Dyspnea: Change at Week 56 (n=4,0) | 0.00 (27.22) | NA (NA) — Data not available as no participant was evaluable.
  Dyspnea: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Dyspnea: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Insomnia: Screening (n=58,31) | 18.39 (28.73) | 18.28 (22.51)
  Insomnia: Change at Week 8 (n=27,16) | 1.23 (25.29) | -8.33 (33.33)
  Insomnia: Change at Week 16 (n=15,7) | 2.22 (32.04) | -4.76 (29.99)
  Insomnia: Change at Week 24 (n=14,1) | -9.52 (46.09) | -33.33 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Insomnia: Change at Week 32 (n=7,2) | 28.57 (23.00) | 16.67 (23.57)
  Insomnia: Change at Week 40 (n=9,1) | 14.81 (24.22) | 33.33 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Insomnia: Change at Week 48 (n=4,1) | 25.00 (31.91) | 33.33 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Insomnia: Change at Week 56 (n=4,0) | 33.33 (27.22) | NA (NA) — Data not available as no participant was evaluable.
  Insomnia: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Insomnia: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Appetite loss: Screening (n=58,31) | 7.47 (19.79) | 5.38 (12.46)
  Appetite loss: Change at Week 8 (n=27,16) | 0.00 (22.65) | -10.42 (23.47)
  Appetite loss: Change at Week 16 (n=15,7) | -2.22 (8.61) | -14.29 (26.23)
  Appetite loss: Change at Week 24 (n=14,1) | -7.14 (19.30) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Appetite loss: Change at Week 32 (n=7,2) | -4.76 (12.60) | 0.00 (0.00)
  Appetite loss: Change at Week 40 (n=9,1) | -7.41 (14.70) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Appetite loss: Change at Week 48 (n=4,1) | -16.67 (19.25) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Appetite loss: Change at Week 56 (n=4,0) | -16.67 (19.25) | NA (NA) — Data not available as no participant was evaluable.
  Appetite loss: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Appetite loss: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Constipation: Screening (n=58,31) | 17.82 (24.36) | 17.20 (25.63)
  Constipation: Change at Week 8 (n=26,16) | 3.85 (25.52) | -4.17 (26.87)
  Constipation: Change at Week 16 (n=15,7) | 4.44 (17.21) | -9.52 (25.20)
  Constipation: Change at Week 24 (n=14,1) | 2.38 (20.52) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Constipation: Change at Week 32 (n=7,2) | -0.00 (38.49) | 16.67 (23.57)
  Constipation: Change at Week 40 (n=9,1) | 3.70 (26.06) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Constipation: Change at Week 48 (n=4,1) | -16.67 (19.25) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Constipation: Change at Week 56 (n=4,0) | 0.00 (27.22) | NA (NA) — Data not available as no participant was evaluable.
  Constipation: Change at Week 64 (n=1,0) | -33.33 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Constipation: Change at Week 72 (n=1,0) | -33.33 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Diarrhea: Screening (n=58,31) | 1.15 (6.14) | 2.15 (8.32)
  Diarrhea: Change at Week 8 (n=27,16) | 0.00 (9.25) | 0.00 (0.00)
  Diarrhea: Change at Week 16 (n=15,7) | -6.67 (18.69) | 0.00 (0.00)
  Diarrhea: Change at Week 24 (n=14,1) | -7.14 (19.30) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Diarrhea: Change at Week 32 (n=7,2) | -4.76 (12.60) | 0.00 (0.00)
  Diarrhea: Change at Week 40 (n=9,1) | 0.00 (0.00) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Diarrhea: Change at Week 48 (n=4,1) | 0.00 (0.00) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Diarrhea: Change at Week 56 (n=4,0) | 0.00 (0.00) | NA (NA) — Data not available as no participant was evaluable.
  Diarrhea: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Diarrhea: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Financial Fn: Screening (n=58,31) | 17.82 (25.91) | 25.81 (34.11)
  Financial Fn: Change at Week 8 (n=27,16) | 6.17 (26.21) | -4.17 (11.39)
  Financial Fn: Change at Week 16 (n=15,7) | 2.22 (15.26) | 9.52 (46.00)
  Financial Fn: Change at Week 24 (n=14,1) | -4.76 (22.10) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Financial Fn: Change at Week 32 (n=7,2) | 0.00 (19.25) | -16.67 (23.57)
  Financial Fn: Change at Week 40 (n=9,1) | -3.70 (26.06) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Financial Fn: Change at Week 48 (n=4,1) | -16.67 (19.25) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable.
  Financial Fn: Change at Week 56 (n=4,0) | -8.33 (31.91) | NA (NA) — Data not available as no participant was evaluable.
  Financial Fn: Change at Week 64 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.
  Financial Fn: Change at Week 72 (n=1,0) | 0.00 (NA) — Standard deviation not available as only 1 participant was evaluable. | NA (NA) — Data not available as no participant was evaluable.

10. Secondary Outcome: Percentage of Participants With Corticosteroid Initiation During the Study Period
Description: Corticosteroid initiation was assessed in participants not receiving corticosteroids at screening. The participant had the event if he/she started on corticosteroids with a dosage greater than equal to (>/=) 2 mg dexamethasone equivalent.
Time Frame: Baseline until recurrence (up to 691 days)
Population: ITT population. Number of participants analyzed signified participants who were not receiving corticosteroids at screening.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 17 | 12
percentage of participants | 58.82 | 41.67

11. Secondary Outcome: Time to Corticosteroid Initiation
Description: Time to corticosteroid initiation was defined as the time from screening to the start date of the first corticosteroid administration in participants not receiving corticosteroids at screening. The participant had the event if he/she started on corticosteroids with a dosage ≥2 mg dexamethasone equivalent. Instead, if the participant was not known to have the event, time was censored at the last available visit date. Time to corticosteroid initiation was estimated using Kaplan Meier method.
Time Frame: Baseline until recurrence (up to 691 days)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 17 | 12
months | 4.49 [1.87 to NA] — The upper limit of 95% confidence interval (CI) was not reached due to higher number (>40%) of censored participants. | 5.93 [0.30 to NA] — The upper limit of 95% confidence interval (CI) was not reached due to higher number (>40%) of censored participants.

12. Secondary Outcome: Percentage of Participants in Each Class of Corticosteroid Use
Description: Corticosteroid use was classified as: 1. No Change (if corticosteroid dose at each assessment was equal to baseline); 2. Decreased (if corticosteroid dose at each assessment was lower than baseline); 3. Increased (corticosteroid dose at each assessment was greater than baseline).
Time Frame: Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, post-treatment follow-up (up to Day 691)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 52 | 28
percentage of participants
  Week 8: Increased (n=52,28) | 17.31 | 17.86
  Week 8: Decreased (n=52,28) | 23.08 | 21.43
  Week 8: No Change (n=52,28) | 59.62 | 60.71
  Week 16: Increased (n=33,18) | 21.21 | 22.22
  Week 16: Decreased (n=33,18) | 36.36 | 27.78
  Week 16: No Change (n=33,18) | 42.42 | 50.00
  Week 24: Increased (n=21,5) | 28.57 | 20.00
  Week 24: Decreased (n=21,5) | 33.33 | 40.00
  Week 24: No Change (n=21,5) | 38.10 | 40.00
  Week 32: Increased (n=14,3) | 14.29 | 33.33
  Week 32: Decreased (n=14,3) | 42.86 | 0.00
  Week 32: No Change (n=14,3) | 42.86 | 66.67
  Week 40: Increased (n=10,2) | 0.00 | 50.00
  Week 40: Decreased (n=10,2) | 60.00 | 0.00
  Week 40: No Change (n=10,2) | 40.00 | 50.00
  Week 48: Increased (n=8,1) | 0.00 | 0.00
  Week 48: Decreased (n=8,1) | 50.00 | 0.00
  Week 48: No Change (n=8,1) | 50.00 | 100.00
  Week 56: Increased (n=6,1) | 0.00 | 0.00
  Week 56: Decreased (n=6,1) | 33.33 | 0.00
  Week 56: No Change (n=6,1) | 66.67 | 100.00
  Week 64: Increased (n=3,1) | 0.00 | 0.00
  Week 64: Decreased (n=3,1) | 0.00 | 0.00
  Week 64: No Change (n=3,1) | 100.00 | 100.00
  Week 72: Increased (n=3,0) | 0.00 | NA — Data not available as no participant was evaluable.
  Week 72: Decreased (n=3,0) | 0.00 | NA — Data not available as no participant was evaluable.
  Week 72: No Change (n=3,0) | 100.00 | NA — Data not available as no participant was evaluable.
  Week 80: Increased (n=1,0) | 0.00 | NA — Data not available as no participant was evaluable.
  Week 80: Decreased (n=1,0) | 0.00 | NA — Data not available as no participant was evaluable.
  Week 80: No Change (n=1,0) | 100.00 | NA — Data not available as no participant was evaluable.
  Week 88: Increased (n=1,0) | 100.00 | NA — Data not available as no participant was evaluable.
  Week 88: Decreased (n=1,0) | 0.00 | NA — Data not available as no participant was evaluable.
  Week 88: No Change (n=1,0) | 0.00 | NA — Data not available as no participant was evaluable.
  Follow-up: Increased (n=9,3) | 33.33 | 0.00
  Follow-up: Decreased (n=9,3) | 0.00 | 33.33
  Follow-up: No Change (n=9,3) | 66.67 | 66.67

13. Secondary Outcome: Percentage of Participants With Karnofsky Performance Status (KPS) Deterioration
Description: Deterioration of KPS was defined as a decrease of at least 20 percentage points with respect to the screening. KPS is an 11-level score which ranges between 0 (death) to 100 (complete healthy status); a higher score represents a higher ability to perform daily tasks.
Time Frame: Baseline until KPS deterioration (up to 691 days)
Population: ITT population. Here, number of participants analyzed signified participants with evaluable data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 37 | 14
percentage of participants | 18.92 | 14.29

14. Secondary Outcome: Time to Karnofsky Performance Status (KPS) Deterioration
Description: Time to KPS deterioration was defined as the time from screening to the first date of deterioration of the KPS score. Deterioration of KPS was defined as a decrease of at least 20 percentage points with respect to the screening. KPS is an 11-level score which ranges between 0 (death) to 100 (complete healthy status); a higher score represents a higher ability to perform daily tasks. Time to KPS deterioration was estimated using Kaplan Meier method. If the participant was not known to have the event, time was censored at the last available visit date.
Time Frame: Baseline until KPS deterioration (up to 691 days)
Population: ITT population. Here, number of participants analyzed signified participants with evaluable data for this outcome.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 37 | 14
months | NA [NA to NA] — Median was not reached as <50% of participants had an event of interest. | NA [NA to NA] — Median was not reached as <50% of participants had an event of interest.

15. Secondary Outcome: Percentage of Participants With World Health Organization (WHO) Performance Status (PS) Deterioration
Description: WHO PS deterioration was defined as a decrease of at least 1 point with respect to the screening value. WHO PS is a 6-level score which ranges between 0 (fully active) to 5 (death); a lower score represents a higher ability to perform daily tasks.
Time Frame: Baseline until WHO PS deterioration (Up to 691 days)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
percentage of participants | 47.46 | 37.50

16. Secondary Outcome: Time to WHO PS Deterioration
Description: Time to WHO PS deterioration was defined as the time from randomization to the first date of deterioration of the WHO performance status score. WHO PS deterioration was defined as a decrease of at least 1 point with respect to the screening value. WHO PS is a 6-level score which ranges between 0 (fully active) to 5 (death); a lower score represents a higher ability to perform daily tasks.
Time Frame: Baseline until WHO PS deterioration (Up to 691 days)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab | Fotemustine
Number analyzed (Participants) | 59 | 32
months | 8.87 [4.17 to NA] — Data could not be estimated as <50% of participants had an event of interest. | NA [NA to NA] — Data could not be estimated as <50% of participants had an event of interest.

ADVERSE EVENTS:
Time Frame: Up to 691 days
Arm/Group | Bevacizumab | Fotemustine
Serious Adverse Events (participants affected / at risk) | 17/59 | 6/32
Other Adverse Events (participants affected / at risk) | 35/59 | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=59) | Fotemustine (N=32)
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 2 | 0
Condition aggravated (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Partial seizures with secondary generalisation (Nervous system disorders) | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=59) | Fotemustine (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 14
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 4
Asthenia (General disorders) | 13 | 4
Fatigue (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 1 | 2
Pyrexia (General disorders) | 5 | 3
Fungal infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 3 | 1
Transaminases increased (Investigations) | 3 | 4
Weight increased (Investigations) | 4 | 1
Convulsion (Nervous system disorders) | 4 | 2
Epilepsy (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 5 | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 3 | 0
Anxiety (Psychiatric disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypertension (Vascular disorders) | 13 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.